CLINICAL TRIAL: NCT03181087
Title: A Phase I, Single-arm, Open Study of the Safety of Umbilical Cord Mesenchymal Stem Cell Local Intramuscular Injection for Treatment of Uterine Scars
Brief Title: Safety of Umbilical Cord Mesenchymal Stem Cell Local Intramuscular Injection for Treatment of Uterine Scars
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The pandemic resulted in no enrollments.
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhengping Liu, MD, Director, Maternal and Child Health Hospital of Foshan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCHHFoshan-1701
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Uterine Scar
Keywords: Mesenchymal Stem Cells; Cesarean Section; Uterine Scar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical cord MSCs Group (Experimental): 1*10^7 Umbilical cord Mesenchymal Stem Cells (MSCs)
  Interventions: Other: Umbilical cord MSCs

INTERVENTIONS:
Other: Umbilical cord MSCs — Participants will receive direct local intramuscular injection of 1*10^7 MSCs (in 1ml of 0.9% saline) in the uterine incision.

SUMMARY:
The purpose of this study is to evaluate the safety of umbilical cord mesenchymal stem cell local intramuscular injection for treatment of uterine scars by a prospective, single-center, open, and single-arm clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women receiving cesarean delivery
* Ages between 21-35 years
* Gestation ages ≥ 37 weeks and < 42 weeks
* Willing to comply with study dosing and completed the entire course of the study
* Willing to give and sign an informed consent form and a photographic release form

Exclusion Criteria:

* Fibroids
* Placenta previa
* Placenta abruption
* Multiple gestation
* Antepartum hemorrhage
* Preeclampsia/Eclampsia
* Hepatic or renal dysfunction
* Any systemic uncontrolled disease
* Inability to provide consent

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-11 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation through vital signs, the results of clinical lab tests and adverse events | 6 months post treatment
  Safety evaluation through vital signs, the results of clinical lab tests and adverse events.

SECONDARY OUTCOMES:
Number of participants with uterine niche | 6 months post treatment
  The niche is defined as a triangular anechoic area at the presumed site of incision in the uterus by transvaginal utrasonography.
Change of uterine scar thickness | 6 weeks, 3 and 6 months post treatment
  The scar thickness be measured using a transvaginal utrasonography
Change of uterine scar area | 6 weeks, 3 and 6 months post treatment
  The scar area will be measured using a transvaginal utrasonography
Number of participants with endometritis | 6 months post treatment
  Endometritis is defined as the presence of at least two of the following signs with no other recognized cause: fever (temperature of at least 38℃), abdominal pain, uterine tenderness, or purulent drainage from the uterus.
Number of participants with wound infection | 6 months post treatment
  Wound infection is defined as the presence of either superficial or deep incisional surgical-site infection characterized by cellulitis or erythema and induration around the incision or purulent discharge from the incision site with or without fever and included necrotizing fasciitis.
Immunoglobulin concentrations in breast milk and serum | 6 weeks, 3 and 6 months post treatment
  Breast milk and serum immunoglobulin (IgG, IgA, IgM) and the complement (C3, C4) are detected by transmission immune turbidity method using automatic biochemical analyzer.
Adverse events occurrence | 6 months post treatment
  Adverse events will be evaluated since the baseline visit until 6 months after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengping Liu, MD, Principal Investigator — Maternal and Child Health Hospital of Foshan
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided